CLINICAL TRIAL: NCT05933330
Title: Hereditary Hemorrhagic Telangiectasia (HHT) and Its Diverse Neurological Manifestations: Unraveling the Intricacies of an Enigmatic Disorder
Brief Title: Hereditary Hemorrhagic Telangiectasia and Neurovascular Manifestations, in the Danish HHT Database
Acronym: DAN-HEMTEL-VM
Status: Active, not recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OP_1656
Record Dates: First submitted 2023-06-15; First posted 2023-07-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic; Intracranial Arteriovenous Malformations
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Danish HHT patient 18-65 years of age
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI — All included patients receive an MRI of the brain

SUMMARY:
With a described prevalence of brain arteriovenous malformations (CAVM) of 12.8% in HHT patients, of whom 10% presents with intracranial hemorrhage, HHT pose a risk of devastating intracranial hemorrhage.

The main objective of the study is to challenge current statements (pros and cons) regarding systematic screening of asymptomatic HHT patients for neurovascular manifestations.

The investigators are thus seeking to answer a question many screening programs have faced.

A screening program should screen for a manageable problem, by a method that is considered cost effective and does not cause negative effect, even when extrapolated to a large cohort. Finally, the positive effect of screening program should outweigh the negative and not cause unnecessary concerns for the patients. The investigators are seeking to draw perspectives from the results to general questions about screening programs.

DETAILED DESCRIPTION:
The Investigators are conducting a study investigating the disease, Hereditary Hemorrhagic Telangiectasia (HHT) and its neuro-logical and -vascular manifestations.

With a described prevalence of brain arteriovenous malformations (CAVM) of 12.8% in HHT patients, of whom 10% presents with intracranial hemorrhage, HHT pose a risk of devastating intracranial hemorrhage.

The main objective of the study is to challenge current statements (pros and cons) regarding systematic screening of asymptomatic HHT patients for neurovascular manifestations.

The investigators seek to fulfill the objective by offering all Danish HHT patients between 18-65 years of age, an MRI of the brain. Participants are asked to answer two questionnaires (SF-36 and BDI II) before and after the MRI. 100 participants are offered an MRI ASL in order, to investigate if this MRI sequence is more suitable to seek out vascular malformations of the brain.

The study is being performed at the University Hospital of Odense; participants receive their MRI at the radiological center closest to their home address. All participants are included, informed, and briefly interviewed over the telephone. Participants will be recruited using the Danish HHT database.

The project consist of 4 main parts.

1. Neurological manifestations of HHT.
2. A screening of all patients in the Danish HHT database, between 18-65 years of age for CAVM.
3. A study of the adverse psychological effect from screening HHT patients in Denmark.
4. An investigation of the optimal screening method for CAVM.

   Part 1

   • Data included in part study 1 is collected retrospectively from the prospectively maintained Danish HHT database.

   Neurological outcomes of all patients in the database, is cross-referenced with the Danish Apoplexy Register (DAP-database), to ensure optimal quality of registered neurological outcomes.

   Part 2
   * Data included in part study 2 is MRI of brain and surgical outcome. The proposed screening method will be conventional MRI, T1, T2 and TOF, of the cerebrum of all HHT patients between 18-65 years of age (n=350). 100 patients will be investigated further with MRI arterial spin labeling (ASL) and included in part 4.

   Part 3 • Data included in part study 3 is SF-36 and BDI II questionaires baseline and 3 months after patients have received an MRI of the brain.

   Part 4 • Data included in part study 4 is MRI of the brain, with comparative ASL sequencing.

   Separated in MRI with conventional sequences compared to MRI with ASL. Data will be reported according to: Reporting standards for angiographic evaluation and endovascular treatment of cerebral arteriovenous malformations, Jayaraman et al. (2011).

   A cost-effectiveness analysis, investigating to prize of an MRI, the cost of additional follow-up of vascular malformations and incidentalomas will be summarized in this part study.

   The data comes from Danish patients with HHT, 18-65 years of age. Continues data is expected to have normal distribution, and will be tested by the shapiro-wilk test.

   In case of normal distribution, oneway anova will be used to test significant levels of difference between the 5 groups (HHT1, HHT2, JP-HHT, Unknown HHT status and not genetically verified).

   If data is not normally distributed Kruskal-Wallis test will be used to test significance.

   Multivariate analyses will be done by logistic regression and in case of non-binary ordered data, ordered logistic regression adjusting for age and gender will be used.

   Dichotomous categorical data will be analyzed of their degree of independence with chi2 test.

   As HHT is inherited autosomal dominantly, and The sample group is only selected by age (18-65 years of age), The investigators expect data to have normal distribution. In case of lack of normal distribution, this could be explained by the fact that HHT is a rare disease with varying penetrance.

   A power analyses for the project shows:

   For the BDI II and SF-36 outcomes with 289 patients a mean change from pre-screening to post-screening could be detected with 80% power if:
   * Pre-post-correlation = 0.5 (assumed to be the lowest realistic value): Change of 0,17 SD could be detected
   * Pre-post-correlation = 0.8 (assumed to be the highest realistic value): Change of 0,10 SD could be detected As a clinical relevant difference typically would be assumed to be at least 0,3 SD, any clinical relevant changes should be detectable with 289 patients.

   A preliminary investigation indicates a 95% inclusion rate (5% of patients does not want to participate, or has already recieved an MRI of brain prior to the study). The investigators expect patients to be less likely to answer the questionnaire send to them 3 months after they have received the results from their brain MRI. Every Friday after initial invitation to the follow-up questionnaire, a reminder will be sent to the patients. after 3 reminders, the patients will finally be called.

   Part 4 - optimal MRI ASL (arterial spin labeling). In order for this study to be successful, The study need at least 10 patients whom have received a brain MRI with ASL that found a Cerebral AVM. In case of lacking case patients, HHT patients who have received an ordinary MRI with angio-sequences, that showed a cerebral AVM will be invited to have an brain MRI with ASL. This examination is done to uncover whether the participants have more cerebral AVM, that is not visible on conventional MRI. previous studies has shown, that roughly, 50% of HHT patients with cerebral AVM has multiple AVMs.

   The Danish HHT center has been situated at Odense University Hospital since 1996 and all HHT patients seen at the center have been included in the national research ´database. In 2015 data were uploaded in a Red Cap database and since then all patients included in the database have received written information and given informed consent. Data regarding date of birth, age, age of diagnosis, HHT type, results of screening for PAVM, CAVM and hepatic AVM (HAVM) are included. Furthermore, data regarding age of debut of epistaxis, results regarding date of neurological events, cerebral ischemia, bleeding, and abscess are also included in the Danish HHT database.

   The study and its part studies, contains personal patient data, and is therefore under the GDPR act.

   The project is approved by the Danish Data Protection Agency and the Region of Southern Denmark´s regional secretariat of Law.

   Data from this project is owned by the Danish HHT-center, and is located at the department of ear, nose and throat surgery at OUH.

   ALL data is only published in anonymized form. Data is only exported from RedCap in pseudononymized form for the purpose of statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* HHT according to the clinical diagnostic criteria (curacao)
* 18-65 years of age.
* registered in the Danish HHT-database

Exclusion Criteria:

* patients has received an MRI of the brain with angio sequences, within the last 5 years.
* contraindications to MRI
* contraindications to self-reported questionnaires (i.e. mental retardation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with HHT (according to the curacao criteria or genetically verified mutations)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of new patients with Cerebral Arteriovenous malformation | 1st of April 2022 - 30th of June 2025.
  MRI verified arteriovenous malformation

SECONDARY OUTCOMES:
Number of new patients with Ischemic stroke | 1st of April 2022 - 30th of June 2025.
  Symptomatic or silent (MRI verified) Ischemic cerebral stroke
Number of new patients with Hemorrhagic stroke | 1st of April 2022 - 30th of June 2025.
  spontaneous CAVM rupture.
Short Form 26 | Baseline - inclusion, and 3 months after screening with MRI, and (in case of treatment) 3 months after treatment. 1st of April 2022 - 30th of June 2025.
  Results from questionnaire SF-36. 0-100. 100 being the best possible.
MRI arterial spin labeling (ASL) | 1st of April 2022 - 30th of June 2025.
  comparison between conventional MRI angio sequences compared to MRI with ASL, in it´s ability to detect CAVM.
Becks Depression Inventory II | Baseline - inclusion, and 3 months after screening with MRI, and (in case of treatment) 3 months after treatment. 1st of April 2022 - 30th of June 2025.
  Results from questionnaire BDI II. 0-61. 61 being the most depressed possible, and 0 the "best".

CONTACTS AND LOCATIONS:
Locations (1):
- Danish HHT-center. Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
All data from the study, will be stored according to danish legislation and GDPR, in certified GDPR servers at OUH, after study completion.